CLINICAL TRIAL: NCT03373214
Title: Randomized, Controlled, Phase 1 Study to Assess Safety and Immunogenicity of Na-GST-1/Alhydrogel®, With or Without a CPG ODN Adjuvant, in Gabonese Adults
Brief Title: Na-GST-1/Alhydrogel With or Without CpG 10104 in Gabonese Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: Centre de Recherche Médicale de Lambaréné (Other); George Washington University (Other); Leiden University Medical Center (Other); Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other); Amsterdam Institute for Global Health and Development (Other)
Responsible Party: Principal Investigator, Maria Elena Bottazzi PhD, Professor, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: HV-03
Record Dates: First submitted 2017-12-06; First posted 2017-12-14 (Actual); Last update posted 2021-01-13 (Actual); Status verified 2021-01

CONDITIONS: Hookworm Infection; Hookworm Disease
Keywords: Human Hookworm; Necator americanus; Hookworm; Hookworm Disease; Iron-deficiency anemia; Soil-transmitted helminth infection; Neglected Tropical Disease; Na-GST-1; CpG
MeSH Terms: conditions — Hookworm Infections; Ancylostomiasis; Anemia, Iron-Deficiency; Neglected Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- 30 µg Na-GST-1 + CPG 10104 (Experimental)
  Interventions: Biological: Na-GST-1; Biological: CPG 10104
- 100 µg Na-GST-1 + CPG 10104 (Experimental)
  Interventions: Biological: Na-GST-1; Biological: CPG 10104
- 100 µg Na-GST-1 (Experimental)
  Interventions: Biological: Na-GST-1

INTERVENTIONS:
Biological: Na-GST-1 — Na-GST-1/Alhydrogel®
Biological: CPG 10104 — CPG 10104
  Arms: 100 µg Na-GST-1 + CPG 10104; 30 µg Na-GST-1 + CPG 10104

SUMMARY:
Na-GST-1 is a protein expressed during the adult stage of the Necator americanus hookworm life cycle that is thought to play a role in the parasite's degradation of host hemoglobin for use as an energy source. Vaccination with recombinant Na-GST-1 has protected dogs and hamsters from infection in challenge studies. This study will evaluate the safety and immunogenicity of administering Na-GST-1 with or without the CpG 10104 immunostimulant to healthy Gabonese adults living in an area of endemic hookworm infection.

DETAILED DESCRIPTION:
Double blind, randomized, controlled, dose-escalation Phase 1 clinical trial in hookworm-exposed adults aged 18 to 50 years living in the area of Lambaréné, Gabon. Participants will receive three doses of the assigned vaccine(s) delivered intramuscularly (deltoid) on approximately Days 0, 56, and 112.

Safety will be measured from the time of each study vaccination (Day 0) through 14 days after each study vaccination by the occurrence of solicited injection site and systemic reactogenicity events.

Unsolicited non-serious adverse events (AEs) will be collected from the time of the first study vaccination through approximately 1 month after each study vaccination. New-onset chronic medical conditions and Serious Adverse Events (SAEs) will be collected from the time of the first study vaccination through approximately 9 months after the final study vaccination (final visit). Clinical laboratory evaluations for safety will be performed on venous blood collected approximately 14 days after each vaccination.

Immunogenicity testing will include IgG antibody responses to each vaccine antigen, by a qualified indirect enzyme-linked immunosorbent assay (ELISA), on serum or plasma obtained prior to each study vaccination and at time points after each vaccination; the functional activity of vaccine-induced antibodies will be assessed by in vitro enzyme neutralization assays.

Recruitment and enrollment into the study will occur on an ongoing basis, with each group being recruited and vaccinated in sequence.

24 subjects will be enrolled into 2 groups:

* Group 1 (n=12):

  * 8 subjects will receive 30 µg Na-GST-1 plus 500 µg CPG 10104 delivered by IM injection in the deltoid muscle
  * 4 subjects will receive 100 µg Na-GST-1 delivered by IM injection in the deltoid muscle
* Group 2 (n=12):

  * 8 subjects will receive 100 µg Na-GST-1 plus 500 µg CPG 10104 delivered by IM injection in the deltoid muscle
  * 4 subjects will receive 100 µg Na-GST-1 delivered by IM injection in the deltoid muscle

ELIGIBILITY:
Inclusion Criteria:

1. Males or females between 18 and 50 years, inclusive, who are long-term residents of the study area.
2. Good general health as determined by means of the screening procedure.
3. Assumed availability for the duration of the trial (13 months).
4. Willingness to participate in the study as evidenced by signing the informed consent document.
5. Negative for hookworm during screening, or if found to be infected with hookworm, has completed a course of three doses of albendazole.

Exclusion Criteria:

1. Pregnancy as determined by a positive urine human choriogonadotropin (hCG) test (if female).
2. Participant unwilling to use reliable contraception up until one month following the final immunization (if female and not surgically sterile, abstinent, at least 2 years post-menopausal, or determined otherwise by medical evaluation to be sterile).
3. Currently lactating and breast-feeding (if female).
4. Inability to correctly answer all questions on the informed consent comprehension questionnaire.
5. Evidence of clinically significant neurologic, cardiac, pulmonary, hepatic, rheumatologic, autoimmune, diabetes, or renal disease by history, physical examination, and/or laboratory studies.
6. Has a diagnosis of schizophrenia, bipolar disease or other major psychiatric condition that would make compliance with study visits/procedures difficult (e.g., subject with psychoses or history of suicide attempt or gesture in the 3 years before study entry, ongoing risk for suicide).
7. Known or suspected immunodeficiency.
8. Laboratory evidence of liver disease (alanine aminotransferase [ALT] greater than 1.25-times the upper reference limit).
9. Laboratory evidence of renal disease (serum creatinine greater than 1.25-times the upper reference limit, or more than 1+ protein, or glucose on urine dipstick testing).
10. Laboratory evidence of hematologic disease (absolute leukocyte count <3500/mm3; absolute leukocyte count >11.0 x 103/mm3; hemoglobin <10.0 g/dl [females] or <12.0 g/dl [males]; or, platelet count <140,000/mm3).
11. Other condition that in the opinion of the investigator could jeopardize the safety or rights of a volunteer participating in the trial or would render them unable to comply with the protocol.
12. Participation in another investigational vaccine or drug trial within 30 days of starting this study or for the duration of the study.
13. History of a severe allergic reaction or anaphylaxis.
14. Severe asthma as defined by the need for daily use of inhalers or emergency room/clinic visit or hospitalization within 6 months of the volunteer's planned first vaccination in the study.
15. Positive for HCV.
16. Positive for HBsAg.
17. Positive for HIV infection.
18. Use of corticosteroids (excluding topical or nasal) or immunosuppressive drugs within 30 days of starting this study or planned use up to one month after the volunteer's final vaccination.
19. Receipt of a live vaccine within past 4 weeks or a killed vaccine within past 2 weeks prior to entry into the study.
20. History of a surgical splenectomy.
21. Receipt of blood products within the 6 months prior to entry into the study.
22. Previous receipt of the Na-GST-1/Alhydrogel® vaccine.
23. Pre-existing autoimmune or antibody-mediated diseases including but not limited to: systemic lupus erythematosus, rheumatoid arthritis, multiple sclerosis, Sjogren's syndrome, autoimmune thrombocytopenia; or laboratory evidence of possible autoimmune disease determined by a positive anti-dsDNA titer, positive rheumatoid factor, proteinuria (greater than trace protein on urine dipstick testing) and/or a positive ANA.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2019-02-28 (Actual); Study Completion 2019-03-30 (Actual)

PRIMARY OUTCOMES:
Vaccine-related Adverse Events | Day 380
  1. To evaluate the safety and reactogenicity of two different dose concentrations of Na-GST-1/Alhydrogel® administered with or without CPG 10104 in healthy Gabonese adults.

SECONDARY OUTCOMES:
Anti-Na-GST-1 IgG Antibody Level on Day 126 | Day 126
  1. To determine the dose/formulation that results in the highest level of anti-Na-GST-1 IgG antibody approximately 14 days after the final vaccination.

OTHER OUTCOMES:
Duration of antibody response to Na-GST-1 | Day 14, 28, 42, 56, 180, 194, 208, 270, 380
  1. To assess and compare the duration of the antibody responses to Na-GST-1 by dose and formulation.
IgG Subclass Distribution to Na-GST-1 | Day 14, 28, 42, 56, 180, 194, 208, 270, 380
  2. To assess the distribution of IgG subclass responses to Na-GST-1 by dose and formulation.

CONTACTS AND LOCATIONS:
Overall Officials: Ayola Adegnika, MD, Principal Investigator — Centre de Recherches Medicales de Lambarené
Locations (1):
- Centre de Récherches Médicales de Lambaréné, Lambaréné, Gabon

IPD SHARING:
Plan to Share IPD: Undecided